CLINICAL TRIAL: NCT02699710
Title: A Phase I, Single Center, Randomized, Open-Label, Study Investigating the Effect of Food, Rabeprazole, Methotrexate and Formulation on the Pharmacokinetics of GDC-0853 and the Effect of GDC-0853 on the Pharmacokinetics of Methotrexate in Healthy Subjects
Brief Title: Effect of Food, Rabeprazole, Methotrexate and Formulation on the Pharmacokinetics (PK) of GDC-0853 and the Effect of GDC-0853 on the PK of Methotrexate in Healthy Subjects
Acronym: QCL117578
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GP29832; 2015-002471-25 (EudraCT Number); QCL117578 (Other: Genentech, Inc.)
Record Dates: First submitted 2016-03-01; First posted 2016-03-04 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Folic Acid; fenebrutinib; Methotrexate; Rabeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: GDC-0853, Rabeprazole (Fasting State) (Experimental): Participants will receive single dose of GDC-0853 (200 milligrams [mg]) in a crossover design as either the capsule or tablet formulation in the fasted state with the final fixed treatment consisting of the tablet formulation administered in the fasted state after prior administration of rabeprazole (20 mg twice daily [BID]) for 3 days.
  Interventions: Drug: GDC-0853; Drug: Rabeprazole
- Part 2: GDC-0853, Rabeprazole (Fasting or Fed State) (Experimental): Participants will receive single dose of GDC-0853 (200 mg) tablet formulation in the fasted or fed state in a crossover design with the final fixed treatment consisting of the tablet formulation administered in the fed state after prior administration of rabeprazole (20 mg BID) for 3 days.
  Interventions: Drug: GDC-0853; Drug: Rabeprazole
- Part 3: GDC-0853, Methotrexate (Experimental): Participants will receive single dose of methotrexate (7.5 mg) under fasting conditions on Day 1 (5 mg folic acid will be administered the following day [Day 2]) and then GDC-0853 (200 mg) tablet formulation twice daily (BID) under fasting conditions (an overnight fast for the morning dose and a 2 hour fast for the evening dose) from Days 15 to 20 after washout period from Days 2 to 14. On Day 21, participants will receive single dose of methotrexate (7.5 mg) with single dose of GDC-0853 (200 mg) tablet formulation under fasting conditions, and folic acid (5 mg) will be administered on Day 22.
  Interventions: Drug: Folic Acid; Drug: GDC-0853; Drug: Methotrexate

INTERVENTIONS:
Drug: Folic Acid — Folic acid will be administered orally as tablet at a single dose of 5 mg.
  Arms: Part 3: GDC-0853, Methotrexate
Drug: GDC-0853 — GDC-0853 will be administered orally as tablet or capsule at a dose of 200 mg.
Drug: Methotrexate — Methotrexate will be administered orally as tablet at a single dose of 7.5 mg.
  Arms: Part 3: GDC-0853, Methotrexate
Drug: Rabeprazole — Rabeprazole will be administered orally as tablet at a dose of 20 mg.
  Arms: Part 1: GDC-0853, Rabeprazole (Fasting State); Part 2: GDC-0853, Rabeprazole (Fasting or Fed State)

SUMMARY:
This study is a Phase I, single center, randomized (Parts 1 and 2 only), open-label, 3 part study. Parts 1 and 2 are 2-way crossover, with 1-fixed sequence, 3-period designs to investigate the effect of formulation, food and rabeprazole on the PK of GDC-0853 in healthy male and female (of non-childbearing potential) participants. Part 3 is a fixed-sequence study with 3 treatments to characterize the steady-state PK of the GDC-0853 tablet; the effect of simultaneous administration of a single dose of methotrexate on the steady-state kinetics of GDC-0853; and the effect of dosing GDC-0853 to steady-state on the single dose PK of methotrexate in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Within body mass index range of 18.0 to 31.0 kilograms per square meter (kg/m^2), inclusive
* For women who are not postmenopausal (greater than or equal to [>/=] 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): these participants will be excluded
* For men: agreement to use a condom plus an additional contraceptive method with their partner during the treatment period and for at least 93 days after the last dose of study drug and agreement to refrain from donating sperm during this same period

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the investigator)
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator
* Participants previously enrolled in this study or participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 90 days prior to Period 1 Check-in (Day -1)
* History of malignancy, except for completely excised basal cell carcinoma or squamous cell carcinoma of the skin or cervical carcinoma in situ
* Female participant is pregnant, lactating or breastfeeding
* Current treatment with medications that are well known to prolong the QT interval
* Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09-03 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

PRIMARY OUTCOMES:
Part 1: Relative Bioavailability of GDC-0853 tablet Compared to GDC-0853 Capsule | Part 1 (Periods 1 to 2 [Period length=5 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Part 1: Area Under the Concentration Time-Curve From Time 0 to Infinity (AUC0-inf) of GDC-0853 Capsule | Part 1 (Periods 1 to 2 [Period length=5 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Part 1: Area Under the Concentration Time-Curve From Time 0 to Last Reported Plasma Concentration (AUC0-t) of GDC-0853 Capsule | Part 1 (Periods 1 to 2 [Period length=5 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Part 1: Maximum Plasma Concentration (Cmax) of GDC-0853 Capsule | Part 1 (Periods 1 to 2 [Period length=5 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Part 1: Time to Maximum Plasma Concentration (Tmax) of GDC-0853 Capsule | Part 1 (Periods 1 to 2 [Period length=5 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Part 1: Apparent half-life (t1/2) of GDC-0853 Capsule | Part 1 (Periods 1 to 2 [Period length=5 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Parts 1 and 2: AUC0-inf of GDC-0853 Tablet | Parts 1 and 2 (Periods 1 to 2 [Period length=5 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Parts 1 and 2: AUC0-t of GDC-0853 Tablet | Parts 1 and 2 (Periods 1 to 2 [Period length=5 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Parts 1 and 2: Cmax of GDC-0853 Tablet | Parts 1 and 2 (Periods 1 to 2 [Period length=5 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Parts 1 and 2: Tmax of GDC-0853 Tablet | Parts 1 and 2 (Periods 1 to 2 [Period length=5 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Parts 1 and 2: Apparent t1/2 of GDC-0853 Tablet | Parts 1 and 2 (Periods 1 to 2 [Period length=5 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Parts 1 and 2: AUC0-inf of GDC-0853 Tablet When Administered With Rabeprazole | Parts 1 and 2 (Period 3 [Period length=8 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Parts 1 and 2: AUC0-t of GDC-0853 Tablet When Administered With Rabeprazole | Parts 1 and 2 (Period 3 [Period length=8 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Parts 1 and 2: Cmax of GDC-0853 Tablet When Administered With Rabeprazole | Parts 1 and 2 (Period 3 [Period length=8 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Parts 1 and 2: Tmax of GDC-0853 Tablet When Administered With Rabeprazole | Parts 1 and 2 (Period 3 [Period length=8 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Parts 1 and 2: Apparent t1/2 of GDC-0853 Tablet When Administered With Rabeprazole | Parts 1 and 2 (Period 3 [Period length=8 days]): Predose (</=1 hour before dosing), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose on Day 1; 24, 36 hours postdose on Day 2; 48 hours postdose on Day 3; 72 hours postdose on Day 4
Part 3: Area Under the Concentration Time-Curve From Time 0 to 24 Hours, Steady State (AUC0-24, ss) of GDC0853 Tablet | Part 3: Predose (</=1 hour before dosing) on Days 17, 18, 19, 20, 21; 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours postdose on Days 20, 21; 16 hours postdose on Day 21; 24 hours postdose on Day 22
Part 3: Maximum Plasma Concentration, Steady State (Cmax, ss) of GDC-0853 Tablet | Part 3: Predose (</=1 hour before dosing) on Days 17, 18, 19, 20, 21; 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours postdose on Days 20, 21; 16 hours postdose on Day 21; 24 hours postdose on Day 22
Part 3: Time to Maximum Plasma Concentration, Steady State (Tmax, ss) of GDC-0853 Tablet | Part 3: Predose (</=1 hour before dosing) on Days 17, 18, 19, 20, 21; 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours postdose on Days 20, 21; 16 hours postdose on Day 21; 24 hours postdose on Day 22
Part 3: Area Under the Concentration Time-Curve From Time 0 to 12 Hours (AUC0-12) of GDC-0853 Tablet When Administered With Methotrexate | Part 3: Predose (</=1 hour before dosing) on Days 17, 18, 19, 20, 21; 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours postdose on Days 20, 21; 16 hours postdose on Day 21; 24 hours postdose on Day 22
Part 3: Cmax of GDC-0853 Tablet When Administered with Methotrexate | Part 3: Predose (</=1 hour before dosing) on Days 17, 18, 19, 20, 21; 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours postdose on Days 20, 21; 16 hours postdose on Day 21; 24 hours postdose on Day 22
Part 3: Tmax of GDC-0853 Tablet When Administered with Methotrexate | Part 3: Predose (</=1 hour before dosing) on Days 17, 18, 19, 20, 21; 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours postdose on Days 20, 21; 16 hours postdose on Day 21; 24 hours postdose on Day 22
Part 3: Area Under the Concentration Time-Curve From Time 0 to 24 Hours (AUC0-24) of Methotrexate When Administered With GDC-0853 | Part 3: Predose (</=1 hour before dosing) on Days 1, 21; 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hours postdose on Days 1, 21; 16 hours postdose on Days 1, 21; 24 hours postdose on Days 2, 22
Part 3: Cmax of Methotrexate When Administered with GDC-0853 Tablet | Part 3: Predose (</=1 hour before dosing) on Days 1, 21; 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 hours postdose on Days 1, 21; 24 hours postdose on Days 2, 22
Part 3: Tmax of Methotrexate When Administered with GDC-0853 Tablet | Part 3: Predose (</=1 hour before dosing) on Days 1, 21; 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 hours postdose on Days 1, 21; 24 hours postdose on Days 2, 22
Part 3: Apparent t1/2 of Methotrexate When Administered With GDC-0853 | Part 3: Predose (</=1 hour before dosing) on Days 1, 21; 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16 hours postdose on Days 1, 21; 24 hours postdose on Days 2, 22

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events | From Baseline up to approximately 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Quotient Clinical Ltd, Clinical Research Unit, Nottingham, United Kingdom